CLINICAL TRIAL: NCT03575819
Title: A Phase 1 Study of FOR46 Administered Every 21 Days in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: A Phase 1 Study of FOR46 in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fortis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FOR46-001
Record Dates: First submitted 2018-06-20; First posted 2018-07-03 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer Metastatic
Keywords: castration-resistant; androgen-signaling blockade progression

STUDY DESIGN:
Intervention Model Description: Following completion of the dose escalation phase of the study and determination of a recommended phase 2 dose, patients will be enrolled into a dose expansion cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FOR46 (Dose Escalation) (Experimental): Eligible patients will receive FOR46 administered as an IV infusion every 21 days. Patients will be enrolled into escalating dose levels during the Dose Escalation period of the study.
  Interventions: Drug: FOR46
- FOR46 (Dose Expansion) (Experimental): Eligible patients will receive FOR46 administered as an IV infusion every 21 days. Patients will receive the maximum tolerated dose during the Dose Expansion period of the study.
  Interventions: Drug: FOR46

INTERVENTIONS:
Drug: FOR46 — FOR46 is an intravenously (IV) administered antibody-drug conjugate (ADC) directed against CD46

SUMMARY:
This study will test the safety and efficacy of FOR46 given every 21 days to patients with metastatic castration-resistant prostate cancer.

The name of the study drug involved in this study is: FOR46 for Injection (FOR46)

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability and antitumor activity of FOR46 in patients with metastatic castration-resistant prostate cancer. This study will be conducted in two parts:

Dose escalation:

This part will evaluate increasing doses of FOR46 to identify the maximum tolerated dose (MTD). The first patient enrolled on the study will receive the lowest dose of FOR46. Once this dose is shown to be safe, a second patient will be enrolled at the next higher dose. Patients will continue to be enrolled into either single or multiple patient groups receiving increasing doses until the MTD is reached.

Dose expansion:

This part of the study will further evaluate the safety, tolerability and antitumor activity of FOR46 at a dose shown to be safe in the dose escalation part of the study. Patients will be enrolled into 1 of 2 groups, based on histology.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years of age
* Has histologically confirmed prostate cancer that is metastatic and has progressed as defined by PCWG3 criteria during or after treatment with at least 1 ASI (eg, abiraterone, enzalutamide, apalutamide), or another second-generation anti-androgen or cytochrome P450 (CYP)17A1 inhibitor, with the most recent ASI administered in the castration-resistant setting
* Has serum testosterone levels < 50 ng/dL during screening. Patients without a history of bilateral orchiectomy are required to remain on luteinizing hormone-releasing hormone (LHRH) analog during the course of protocol therapy
* ECOG performance status of 0 or 1
* Adequate hematologic, renal and hepatic function
* Males with female partners of childbearing potential must agree to use 2 effective methods of contraception
* Patients must provide signed informed consent
* Patients enrolled into the dose expansion phase must have prostate carcinoma without histologic evidence of small-cell/neuroendocrine carcinoma features on prior biopsy or must have unequivocal histologic evidence of small-cell/neuroendocrine prostate carcinoma (pure or mixed). Patients with treatment-emergent small-cell neuroendocrine cancer (pure or mixed) may have received no more than on prior chemotherapy regimen for mCRPC
* Patients enrolled into the dose expansion phase must be willing to undergo a metastatic tumor biopsy or has tissue available from a prior post-castration resistant tumor biopsy

Exclusion Criteria:

* Persistent clinically significant toxicities from previous anticancer therapy
* Has NCI CTCAE Grade ≥ 2 peripheral neuropathy from any etiology or has a genetic disorder that is associated with peripheral neuropathy even without current neuropathic manifestations
* Prior treatment with cytotoxic chemotherapy for mCRPC (chemotherapy in the hormone-sensitive setting is allowed if > 6 months before study entry)
* Has received external-beam radiation or systemic anticancer therapy within 14 days before first dose of FOR46
* Has received treatment with an investigational drug within 28 days before first dose of FOR46
* Has had a major surgical procedure within 28 days before administration of FOR46 dose
* Clinically significant cardiovascular disease
* Uncontrolled, clinically significant pulmonary disease
* Has a history of brain or leptomeningeal metastases.
* Uncontrolled intercurrent illness
* Has a known positive status for HIV or either active/chronic hepatitis B/C
* Requires medications that are strong inhibitors or strong inducers of CYP3A4
* [Dose escalation only] Has a history of episodic atrial fibrillation or flutter (patients with chronic atrial fibrillation are not excluded)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Occurrence of toxicity | Through 1 month following last dose
  Type, incidence, severity, seriousness, and relatedness of adverse events.
Occurrence of dose-limiting toxicities | Through 1 month following last dose
  The severity and incidence of dose-limiting toxicities related to escalating dose levels of FOR46
Disease response/composite response | 12 months
  Decline in serum prostate-specific antigen greater than 50% from baseline, confirmed by repeat measurement and objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Characterize FOR46 plasma concentration | Through 1 month following last dose
  FOR46 maximum plasma concentration
Characterize the FOR46 area under the curve | Through 1 month following last dose
  FOR46 area under the plasma concentration-time curve
Characterize FOR46 elimination | Through 1 month following last dose
  FOR46 elimination half-life
Antidrug Antibodies | Through 1 month following last dose
  Change from baseline in serum levels of antidrug antibodies
Median radiographic progression-free survival | 12 months
  Assessed by Prostate Cancer Clinical Trials Working Group 3 criteria

OTHER OUTCOMES:
Exploratory Endpoint: Tumor expression of CD46 | Through 1 month following last dose
  Association between level of tumor expression of CD46 by immunohistochemistry (IHC) analysis with clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dorr, MD, Study Director — Fortis Therapeutics, Inc.
Locations (5):
- United States (5):
  - UCLA Institute of Urologic Oncology, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - OHSU Knight Cancer Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aggarwal RR, Vuky J, VanderWeele D, Rettig M, Heath EI, Quigley D, Huang J, Chumber A, Cheung A, Foye A, Leung S, Abbey J, Dorr A, Nasoff M, Hunter J, Wang S, Flavell RR, Fong L, Liu B, Small EJ. Phase I, First-in-Human Study of FOR46 (FG-3246), an Immune-Modulating Antibody-Drug Conjugate Targeting CD46, in Patients With Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2025 May 20;43(15):1824-1834. doi: 10.1200/JCO-24-01989. Epub 2025 Mar 26. PMID 40138611